CLINICAL TRIAL: NCT04604379
Title: A Multicentre, Non-interventional Retrospective Study of Treatment Outcomes From Treatment With Dysport ® (Clostridium Botulinum Type A Toxin-haemagglutinin Complex, Abobotulinumtoxin-A) Injections in Adults for Upper and/or Lower Limb Focal Spasticity in Real-world Clinical Practice in the United Kingdom
Brief Title: A Study to Review Treatment Outcomes From Treatment With Dysport® Injections in Adults for Upper and/or Lower Limb Focal Spasticity
Acronym: DYSCOVER
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-GB-52120-277
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Upper and/or Lower Limb Focal Spasticity
Keywords: Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this retrospective study is to describe the real-world outcomes with the treatment of adult patients with Dysport® injections for focal upper limb spasticity (ULS) and/or focal lower limb spasticity (LLS) in NHS hospital settings in the United Kingdom (UK).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with focal ULS and/or LLS for whom aboBoNT-A (Dysport®) was prescribed in line with the SmPC (according to clinician judgement).
* Patients initiated on aboBoNT-A for focal ULS after the 31st January 2016 and/or for focal LLS after the 06th December 2016.
* Patients receiving ≥1 injection(s) (i.e. ≥1 treatment cycle) of aboBoNT-A during the observation period, in line with Dysport® Summary of Product Characteristics (SmPC).
* Patients aged ≥18 years old at the time of the first aboBoNT-A injection for focal ULS and/or LLS.
* Patient is naïve to treatment with any type of BoNT-A during the 6 months prior to initiation of aboBoNT-A.
* Patients treated at the participating centre for the duration of the observation period, with data recorded in the medical records available for review.

Exclusion Criteria:

* Patients with an interval of <12 weeks between aboBoNT-A treatments
* Patients are participating (or who have participated) in an interventional clinical trial of an investigational medicinal product indicated for spasticity which may influence and confound the real-world data collected for this study.
* Patients treated with aboBoNT-A off-license, this may include off-license indications, muscles indicated for injection or dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3-5 Secondary care centres in the UK
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Average total dose of AboBoNT-A for focal upper limb and/or lower limb spasticity per treatment session | From baseline (when each patient received their first treatment) to 52 weeks (±6 weeks) post baseline
Average interval between AboBoNT-A injections throughout the observation period for focal ULS and/or LLS | From baseline to 52 weeks (±6 weeks) post baseline

SECONDARY OUTCOMES:
Average age at diagnosis of neurological condition | Baseline
Average age at first AboBoNT-A injection | Baseline
Average age at diagnosis of spasticity | Baseline
Sex distribution (Male, Female) | Baseline
Presence of underlying neurological condition: stroke, injury, chronic disease (multiple sclerosis, other) | Baseline
Presence of location of spasticity (specify: right lower limb, left lower limb, right upper limb, left upper limb, unilateral, bilateral spasticity for lower and upper limb) | Baseline
  Data collected at index date up to 6 weeks prior to index date (when each patient received their first treatment)
Presence of previous spasticity-related treatments ongoing at index event, if available: antispasticity medications, pain medications and opioids, neurolytic agent, surgery, physiotherapy and occupational therapy | Baseline
Presence of comorbidities: bowel conditions (irritable bowel syndrome, irritable bowel disease), urinary tract infections, chest infections, anxiety or depression, alcohol dependence/substance abuse. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (3):
- United Kingdom (3):
  - Kings College Hospital, London
  - Colman Hospital, Norwich
  - York Hospital, York